CLINICAL TRIAL: NCT05319574
Title: Preoperative Stereotactic Body Radiotherapy and Platinum-based Doublet Chemotherapy Plus Tislelizumab (Immunotherapy) for Operable Stage II to III EGFR Wild-type Non-small Cell Lung Cancer
Brief Title: SBRT Followed by Neoadjuvant Immunochemotherapy in Resectable Stage II to III Non-small Cell Lung Cancer
Acronym: SACTION01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Hong, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC B2022-159-01
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non small cell lung cancer; Neoadjuvant; Immunotherapy; SBRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant SBRT plus immunochemotherapy (Experimental): Stereotactic body radiation therapy (8Gy*3d) followed by Tislelizumab (200mg) with platinum-based doublet chemotherapy administered pre-operatively every 3 weeks for 2 cycles before surgical resection
  Interventions: Radiation: SBRT; Drug: Tislelizumab

INTERVENTIONS:
Radiation: SBRT — Stereotactic body radiation therapy delivered with a fixed dose (8Gy) in 3 daily fractions 1-7 days before the first cycle of immunochemotherapy
  Other Names: stereotactic body radiation therapy
Drug: Tislelizumab — 200mg q3w for two cycles administrated concurrently with chemotherapy

SUMMARY:
The purpose of this study is to find out the effectiveness stereotactic body radiation therapy (SBRT) followed by two cycles of Tislelizumab (PD-1 inhibitor) with chemotherapy as treatment for operable stage II to III non-small cell lung cancer (NSCLC) prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically or cytologically proven clinical stages II and III NSCLC (according to the 8th AJCC edition) and is considered eligible for surgical resection with curative intent. Besides, T3-4N2 stage IIIB disease deemed potentially resectable by MDT group is also allowed.
2. Measureable disease, as defined by RECIST v1.1.
3. Written informed consent and HIPAA obtained from the subject prior to performing any protocol-related procedures.
4. EGFR mutational status should be tested in all non-squamous carcinoma, and only patients with non-EGFR-TKI sensitizing mutation (19del or L858R) are allowed. For squamous cell carcinoma, EGFR mutational test is not required.
5. Age > 18 years at time of study entry
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT), and alkaline phosphatase ≤ 2.5 x institutional upper limit of normal (ULN).
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
8. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

   Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
9. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
10. No prior therapy for their lung cancer.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3 weeks.
2. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ, in-situ urinary bladder cancer , treated localized prostate cancer and ductal carcinoma-in situ.
   * Indolent hematological malignancies
3. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal,inhaled, topical steroids, or local steroid injections (e.g., intra articular injection), corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, and steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
4. Any unresolved toxicity (CTCAE grade 2) from therapy for a prior malignancy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy).
5. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
6. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). No active diverticulitis within the previous 3 months. The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
7. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
8. History of active primary immunodeficiency.
9. History of allogeneic organ transplant.
10. History of hypersensitivity to tislelizumab or any excipient.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
12. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
13. History of leptomeningeal carcinomatosis.
14. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
15. Subjects with uncontrolled seizures.
16. History of interstitial lung disease, idiopathic pulmonary fibrosis, pneumonitis (including drug induced), or evidence of active pneumonitis on screening chest CT scan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-04-24 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | From date of enrollment until one month after resection
  MPR is defined as ≤10% residual viable tumor in the resected specimen

SECONDARY OUTCOMES:
Pathologic Complete response (PCR) | From date of enrollment until one month after resection
  PCR is defined as no residual viable tumor in the resected specimen
Resected rate | From date of enrollment to an average of 18 weeks after the first dose
  Resected rate is defined as the percentage of patients that undergo surgical resection after neoadjuvant treatment
Disease-free survival | From date of SBRT start date until the date of first documented progression or date of death from any cause, whichever came first, assessed every 6 months for 2 years , then yearly thereafter till year 5
  Disease recurrence or death from any cause assessed using history, physical examination and CT scanning, histologically or cytologically confirmed whenever possible

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhao ZR, Liu SL, Zhou T, Chen G, Long H, Su XD, Zhang X, Fu JH, Lin P, Zhang LJ, Rong TH, Wu JD, Li ZC, Su HL, Chen JY, Yang YP, Lin YB, Xi M, Yang H. Stereotactic body radiotherapy with sequential tislelizumab and chemotherapy as neoadjuvant therapy in patients with resectable non-small-cell lung cancer in China (SACTION01): a single-arm, single-centre, phase 2 trial. Lancet Respir Med. 2024 Dec;12(12):988-996. doi: 10.1016/S2213-2600(24)00215-7. Epub 2024 Sep 18. PMID 39305910